CLINICAL TRIAL: NCT03482765
Title: A Double-blind Randomized, Placebo-controlled, Parallel Group Study of the Efficacy and Safety of Probiotics (UABla-12™ and DDS®-1) on Digestive Health in IBS Subjects
Brief Title: A Study of Probiotics in IBS Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UAS/170901/PB/IBS
Record Dates: First submitted 2018-02-22; First posted 2018-03-29 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: IBS
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Apart from the participant and Investigator, the study team is also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic 1 (Experimental): Probiotic 1: A dietary probiotic supplement which contains Bifidobacterium lactis. Dose: > 10 billion CFU, Frequency: 1 capsule/day, duration: 6 weeks.
  Interventions: Dietary Supplement: Probiotic 1
- Probiotic 2 (Experimental): Probiotic 2: A dietary probiotic supplement which contains Lactobacillus acidophilus. Dose: > 10 billion CFU, Frequency: 1 capsule/day, duration: 6 weeks.
  Interventions: Dietary Supplement: Probiotic 2
- Placebo (Placebo Comparator): The Placebo contains MCC.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic 1 — The product under investigation is a unique probiotic.
  Other Names: Bifidobacterium lactis
  Arms: Probiotic 1
Dietary Supplement: Probiotic 2 — The product under investigation is a unique probiotic.
  Other Names: Lactobacillus acidophilus
  Arms: Probiotic 2
Other: Placebo — Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
For the current study, the primary outcome is to evaluate the effect of IP on abdominal pain.

The secondary outcome is to assess the effect of IP on IBS-Symptom Severity, IBS-related quality of life, stool form and consistency and on mental status.

Thus providing an effective objective in improving the gut health and symptomatic relief in IBS patients.

DETAILED DESCRIPTION:
This study aims to determine the effect of probiotics, as the investigational products (IPs) in subjects satisfying the Rome IV criteria for IBS. Three hundred and sixty six subjects between 18 to 70 years of age and with a positive diagnosis of Rome IV IBS criteria (IBS-C, D, M and U types) and moderate to severe abdominal pain intensity will be recruited in a multi-center, double-blind, parallel group, placebo-controlled randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Literate (as defined by the basic capability to read and understand in the languages approved for the study), male and female subjects in age range of 18-70 years.
* Presence of Rome IV diagnostic criteria for IBS.

Exclusion Criteria:

* Anemic subjects with Hb < 10 g/dl.
* Subjects with organic disease (to be ruled out by physician based on prior history and physical examination).
* Subjects with a history of surgical resection of the stomach, small intestine or large intestine.
* Subjects with a history of or complications from inflammatory bowel disease (Crohn's disease or ulcerative colitis) and ischemic colitis.
* Subjects with complications from infectious enteritis, hyperthyroidism or hypothyroidism.
* Subjects with a history of any diet-based intolerance (gluten or lactose intolerance).
* Subjects with a history of drug or alcohol abuse within the past 6 months.
* Subjects with a history of or complications from malignant tumors.
* Subjects with severe depression or an anxiety disorder, which could potentially affect the efficacy evaluation (as determined by the qualified investigator).
* Subjects with uncontrolled hypertension (≥140/90 mm Hg).
* Subjects with complications from serious cardiovascular diseases, respiratory diseases, endocrinological and gynecological disorder, renal diseases, hepatic diseases, gastrointestinal diseases (excluding IBS), blood diseases or neurological or psychiatric diseases.
* Subjects who are pregnant, breastfeeding or planning on becoming pregnant throughout the course of the study.
* Subjects with a history of dysmenorrhea.
* Subjects with any unstable medical conditions.
* Subjects with uncontrolled Type II diabetes mellitus.
* Subjects with a history of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years after diagnosis are acceptable.
* Subjects who are immuno-compromised (HIV positive, on anti-rejection medication, rheumatoid arthritis).
* Subjects with any medical condition or a history of abdominal surgery that is deemed exclusionary by the qualified investigator.
* Subjects with an active eating disorder.
* Subjects who have used an over-the-counter or prescription laxative medication or any other herbal agents affecting GI motility within 2 weeks prior to screening.
* Subjects who have used probiotic or fiber supplements (or probiotic/fiber enriched foods) or an antibiotic within 4 weeks prior to screening.
* Subjects who have used IBS specific treatments within 4 weeks prior to screening.
* Subjects who currently consume greater than 2 standard alcoholic drinks per day from past 3 months.
* Subjects who smoke ≥ 1 cigarette per day. Occasional (Non-daily) smokers will be allowed.
* Subjects who have participated in a clinical research trial within 30 days prior to randomization.
* Subjects with an allergy or sensitivity to the probiotic products.
* Subjects who are cognitively impaired and/or who are unable to give an informed consent.
* Subjects who have abnormal laboratory results or any other medical or psychological condition which, in the opinion of the qualified investigator, may adversely affect the subjects' ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in abdominal pain severity | 42 days
  The change at Day 42 will be assessed by subject dairy.

SECONDARY OUTCOMES:
Change in abdominal pain severity | Day 21
  The change at Day 21 will be assessed by subject dairy
Change in IBS symptoms | Day 42
  The change at Day 42 will be compared to baseline
Change in stool consistency | Day 42
  The change at Day 42 will be compared to baseline by specific questionnaire
Change in Quality of Life | Day 42
  The change at Day 42 will be compared to baseline by specific questionnaire
Change in daily number of stools | Day 42
  The change at Day 42 will be compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Srivastava, M.D., Study Director — Vedic Lifesciences
Locations (12):
- India (12):
  - Apex Gastro Clinic, Ahmedabad, Gujarat
  - Gastrocare & Liver Clinic, Ahmedabad, Gujarat
  - The Gut Clinic, Mumbai, Maharashtra
  - Vazifdar Clinic, Mumbai, Maharashtra
  - Stress Test Clinic, Mumbai, Maharashtra
  - Shantaee Nursing Home, Mumbai, Maharashtra
  - Dr Sanjeev Khanna's Clinic, Mumbai, Maharashtra
  - Ameeta Nursing home, Mumbai, Maharashtra
  - Lancelot Kidney and GI Center, Mumbai, Maharashtra
  - Kshirsagar Nursing Home, Mumbai, Maharashtra
  - Samarth Clinic, Navi Mumbai, Maharashtra
  - Sampada Hospital, Thane, Maharashtra